CLINICAL TRIAL: NCT00804947
Title: Ensayo Fase II de Trasplante autólogo de Sangre periférica en Pacientes Con Mieloma múltiple Tras Acondicionamiento Con Busulfan Intravenoso y Melfalan
Brief Title: Autologous Stem Cell Transplant (ASCT) With Intravenous Busulfan and Melphalan as Conditioning Regimen
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: Javier de la Rubia, Hematology Service. Hospital La Fe. Valencia, Spain
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BuMel-MM
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Multiple Myeloma
Keywords: Autologous transplantation; Multiple Myeloma; Intravenous Busulfan
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous busulfan and melphalan (Experimental)
  Interventions: Drug: Intravenous busulfan and melphalan

INTERVENTIONS:
Drug: Intravenous busulfan and melphalan — BU is administered intravenously at a dose of 3.2 mg/kg over three hours once a day on days -5 to -3 (total dose 9.6 mg/kg), followed by MEL at a dose of 140 mg/m2 on day -2. After one day of rest, progenitor cells are infused on day 0.

SUMMARY:
Analyze the results of ASCT using intravenous Busulfan and Melphalan as conditioning regimen for patients with Multiple Myeloma.

DETAILED DESCRIPTION:
Primary Efficacy and safety of the procedure in terms of number of remissions, survival, event-free survival, relapse risk, and early transplant-related mortality (up to day +100).

Secondary Graft kinetics (time to neutrophil and platelet recovery after ASCT) 2.Analyze the presence of transplant-related complications (infections, sinusoidal occlusive syndrome and others) 3.Analyze prognostic factors for engraftment, remission rate, relapse risk, disease-free and overall survival after ASCT

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma
* Male or female subject age >= 70 years
* The subject has received at least one previous line of therapy including:
* Front-line treatment with VBMCP/VBAD or VAD or second-line therapy with regimens including bortezomib, thalidomide or lenalidomide
* The subject has given voluntary written informed consent

Exclusion Criteria:

* Use of bortezomib, thalidomide or lenalidomide as front-line therapy
* ECOG satus >=2
* Left ventricular ejection fraction <40%
* DLCO and FVC <39% theoretical value
* Abnormal liver function(total bilirubin > 2 mg/dL and/or ALT or AST > 3 x ULN)
* Serum creatinine at transplant >1.6 mg/dL and/or creatinine clearance < 65 mL/minute
* Subject has an active systemic infection requiring treatment
* Subject had a myocardial infarction within 6 months of enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrythmias
* Subject has any other serious medical condition (severe hepatic impairment, pericardial disease, acute diffuse infiltrative pulmonary disease) or psychiatric illness that could potentially interfere with the completion of treatment of this protocol
* Subject is known to be immunodeficiency virus (HIV)-positive
* Subject has received an experimental drug or used and experimental medical device within 4 weeks before enrollment
* If female, the subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative pregnancy test at screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to analyze the safety profile and determine the overall response rate after ASCT with this conditioning regimen. | Within the first three months after transplant

SECONDARY OUTCOMES:
Evaluate the complete response (CR) rate, the duration of the response, time to progression, event-free and overall survival | Up to 5 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A Sanz, MD, Study Director — S: de Hematología. Hospital La Fe, Valencia. Spain
Locations (6):
- Spain (6):
  - Hospital Insular Canarias, Las Palmas de Gran Canaria, Las Palmas
  - H La Princesa, Madrid, Madrid
  - H. 12 de Octubre, Madrid, Madrid
  - S. de Hematología. Hospital La Fe, Valencia, Valencia
  - Hospital Clínico, Valencia, Valencia
  - Hospital Dr. Peset, Valencia, Valencia

REFERENCES:
- [Derived] Blanes M, Lahuerta JJ, Gonzalez JD, Ribas P, Solano C, Alegre A, Blade J, San Miguel JF, Sanz MA, de la Rubia J. Intravenous busulfan and melphalan as a conditioning regimen for autologous stem cell transplantation in patients with newly diagnosed multiple myeloma: a matched comparison to a melphalan-only approach. Biol Blood Marrow Transplant. 2013 Jan;19(1):69-74. doi: 10.1016/j.bbmt.2012.08.009. Epub 2012 Aug 13. PMID 22897964